CLINICAL TRIAL: NCT03983694
Title: Cerebral Haemodynamic Changes by Red Blood Cell Transfusion in Neonates
Status: Completed | Type: Observational
Sponsor: Gorm Greisen (Other)
Collaborators: Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other)
Responsible Party: Sponsor-Investigator, Gorm Greisen, professor, Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Other Study IDs: BabyLux transfusion
Record Dates: First submitted 2019-06-07; First posted 2019-06-12 (Actual); Last update posted 2023-03-28 (Actual); Status verified 2023-03

CONDITIONS: Cerebral Haemodynamics; Erythrocyte Transfusion
MeSH Terms: interventions — Erythrocyte Transfusion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- BabyLux device: Cerebral haemodynamics of neonates undergoing erythrocyte transfusion according to the local clinical guidelines are monitored with BabyLux device before and after transfusion and with traditional NIRS during itself.
  Interventions: Other: Erythrocyte transfusion

INTERVENTIONS:
Other: Erythrocyte transfusion — The cerebro-vascular effects of a clinically prescribed erytrocyte (red blood cell) transfusion is examined. Before the transfusion, BabyLux sensor is placed on the neonatal fronto-parietal region and held in place by a self-adhesive bandage. A baseline prior to transfusion is established through a series of five repeated measurements of 1 minute taken during a stable period just before the transfusion is started. Once transfusion has ended, another series of five repeated measurements of 1 minute taken during a stable period are performed to determine the responses. Cerebral oxygenation as determined by a commercial spatially resolved NIRS device with neonatal sensor will be continuously recorded during transfusion.

SUMMARY:
The timing and the indications for red blood cell (RBC) transfusions remain one of the most controversial topic in Neonatology. Indeed, biomarkers routinely used to discriminate between patients that will benefit from RBC transfusion appear insufficient. Tissue oxygenation could be useful to determine the need for transfusion.

This study aims to assess the effects of RBC transfusion on cerebral haemodynamics and oxygenation in neonates with a new hybrid optical device (BabyLux) integrating time-resolved spectroscopy (NIRS-TRS) and diffuse correlation spectroscopy (DCS).

It is hypothesized that cerebral blood flow decreases after RBC transfusion, whereas cerebral oxygenation and oxygen metabolism are unchanged.

DETAILED DESCRIPTION:
The BabyLux hybrid setup can determine the following parameters in the same tissue sample non-invasively and continuously with a high temporal resolution (0.1-0.2 Hz):

* Cerebral blood flow index (CBFi), i.e. an index that is proportional with CBF
* Concentration of oxyhaemoglobin (O2Hb)
* Concentration of deoxyhaemoglobin (dHb)
* Total haemoglobin concentration (tHb)
* Tissue oxygen saturation (rStO2)
* Cerebral metabolic rate of oxygen index (CMRO2i), i.e. an index that is proportional with CMRO2 Hence, the BabyLux device allows assessment of key parameters of cerebral haemodynamics and, in particular, to examine if the percentage change of cerebral metabolic rate for oxygen is close to the expected zero, as an external quality control of the separate NIRS parameters.

There are no studies on RBC transfusion in neonates evaluating cerebral haemodynamic utilizing DCS and TRS combined.

Hence, primary aim of this study is:

- to assess the effect of RBC transfusion on cerebral haemodynamics and oxygenation as measured by the Babylux device.

Secondary aims are:

* to quantify the effect of estimated ∆[Hb] on the differential path length factor (DPF);
* to compare two different NIRS devices and techniques. BabyLux measurement will be performed before and after RBC transfusion, whereas during RBC transfusion cerebral oxygenation will be monitored with a spatially resolved continuous wave (CW) NIRS.

ELIGIBILITY:
Inclusion Criteria:

* RBC transfusion prescribed according to local NICU guidelines
* Corrected age < 4 weeks corrected age
* Signed informed consent

Exclusion Criteria:

None

Ages: 0 Weeks to 4 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Newborn infants admitted to a neonatal intensive care unit and who need an erythrocyte transfusion
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2019-06-20 (Actual); Primary Completion 2022-07-31 (Actual); Study Completion 2022-12-20 (Actual)

PRIMARY OUTCOMES:
Cerebral metabolic rate of oxygen index (CMRO2i) | From immediately before to immediately after RBC transfusion
  The change in an index proportional to CMRO2

SECONDARY OUTCOMES:
Tissue oxygen saturation (rStO2) | From immediately before to immediately after RBC transfusion
  The change in oxygenated haemoglobin/total haemoglobin
Cerebral blood flow index (CBFi) | From immediately before to immediately after RBC transfusion
  The change in an index proportional to CBF
Differential path length factor (DPF) | From immediately before to immediately after RBC transfusion
  The change in an optical parameter for physiological measurement using NIRS

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione IRCCS Ca' Granda, Milan, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Banerjee J, Aladangady N. Biomarkers to decide red blood cell transfusion in newborn infants. Transfusion. 2014 Oct;54(10):2574-82. doi: 10.1111/trf.12670. Epub 2014 May 5. PMID 24797124
- [Background] Cerussi A, Van Woerkom R, Waffarn F, Tromberg B. Noninvasive monitoring of red blood cell transfusion in very low birthweight infants using diffuse optical spectroscopy. J Biomed Opt. 2005 Sep-Oct;10(5):051401. doi: 10.1117/1.2080102. PMID 16292938
- [Background] Koyano K, Kusaka T, Nakamura S, Nakamura M, Konishi Y, Miki T, Ueno M, Yasuda S, Okada H, Nishida T, Isobe K, Itoh S. The effect of blood transfusion on cerebral hemodynamics in preterm infants. Transfusion. 2013 Jul;53(7):1459-67. doi: 10.1111/j.1537-2995.2012.03953.x. Epub 2012 Nov 12. PMID 23145971
- [Background] Bailey SM, Hendricks-Munoz KD, Wells JT, Mally P. Packed red blood cell transfusion increases regional cerebral and splanchnic tissue oxygen saturation in anemic symptomatic preterm infants. Am J Perinatol. 2010 Jun;27(6):445-53. doi: 10.1055/s-0030-1247598. Epub 2010 Jan 22. PMID 20099219
- [Background] Dani C, Pratesi S, Fontanelli G, Barp J, Bertini G. Blood transfusions increase cerebral, splanchnic, and renal oxygenation in anemic preterm infants. Transfusion. 2010 Jun;50(6):1220-6. doi: 10.1111/j.1537-2995.2009.02575.x. Epub 2010 Jan 22. PMID 20113454
- [Background] Sandal G, Oguz SS, Erdeve O, Akar M, Uras N, Dilmen U. Assessment of red blood cell transfusion and transfusion duration on cerebral and mesenteric oxygenation using near-infrared spectroscopy in preterm infants with symptomatic anemia. Transfusion. 2014 Apr;54(4):1100-5. doi: 10.1111/trf.12359. Epub 2013 Jul 31. PMID 23901886
- See also: The BabyLux project web-site — http://www.babylux-project.eu/